CLINICAL TRIAL: NCT04094142
Title: Phase II Trial of Acalabrutinib With Rituximab and Lenalidomide in Relapsed/Refractory B-cell Non-Hodgkin Lymphoma
Brief Title: Acalabrutinib With Rituximab and Lenalidomide in Relapsed/Refractory B-cell Non-Hodgkin Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, YOUNGIL KOH, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1811-092-988
Record Dates: First submitted 2019-07-19; First posted 2019-09-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Non-hodgkin Lymphoma,B Cell
MeSH Terms: interventions — acalabrutinib; Lenalidomide; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment arm (Experimental): Acalabrutinib is provided as hard gelatin capsules for oral administration. Acalabrutinib 100 mg will be administered approximately every 12 hours from day 1 to day 28 Rituximab is provided as single-use vials for intravenous administration only. Rituximab 375 mg/m2 will be administered on day 1.
  Lenalidomide is provided as opaque hard capsules for oral administration. Lenalidomide 20 mg will be administered once daily from day 1 to day 21
  Interventions: Drug: Acalabrutinib

INTERVENTIONS:
Drug: Acalabrutinib — Acalabrutinib, lenalidomide, rituximab will be given as described in the "Arms" decriptions. Day 1 to day 28 is considered one cycle, and cycles will be repeated every 4-weeks, for 6 cycles.
  After 6 cycles, maintenance of acalabrutinib 100mg bid will be administered up to 1 year for subjects whose best responses- to the regimen are partial response or complete remission.
  Other Names: Lenalidomide; Rituximab

SUMMARY:
NCCN guidelines for B cell lymphoma suggest that patients with relapsed/refractory aggressive NHL who are candidate for high-dose therapy should receive combination of cytotoxic chemotherapies as 2nd line treatment. However, proportion of patients who are adequately salvaged by second line chemotherapy and high-dose chemotherapy with stem cell rescue is unsatisfactory. Moreover, many fragile patients are unfit for salvage cytotoxic chemotherapy and/or high-dose chemotherapy. Hence, most of patients with relapsed/refractory aggressive B-cell NHL is ultimately candidate for less-cytotoxic drugs with targeted approach. This trial is phase II trial of acalabrutinib in combination with rituximab and lenalidomide for these patients.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women ≥ 18 years of age.
2. Diagnosed with aggressive B cell non-Hodgkin lymphoma

   * Diffuse large B cell lymphoma (Both GCB and non-GCB)

     : GCB type should not be more than 40% (N=26) of whole study population (Would limit number of GCB patients by maximum of 26)
   * Primary mediastinal B cell lymphoma
   * Transformed follicular lymphoma
   * Small lymphocytic lymphoma with Richter transformation
3. Failed previous treatments and last dose administered must be more than 2-week ahead from enrollment

   * Should have received anti-CD20 based chemotherapy previously
   * Failed at least two lines of therapy if patient is candidate for autologous stem cell transplantation
   * Failed frontline therapy if patient is ineligible for autologous stem cell transplantation
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2
5. Woman of childbearing potential (WOCBP) who are sexually active must have 2 negative urine hCG test prior to first dose, then every week for the first month of study period, then every 4 weeks afterwards during treatment period if menses are regular or every 2 weeks if menses are irregular. Urine hCG test must be done 4 weeks after the last dose of acalabrutinib, lenalidomide and rituximab. WOCBP must use 2 methods including at least 1 highly effective method of contraception for 4 weeks prior to first dose, during treatment period and for 4 weeks after the last dose of acalabrutinib, lenalidomide and for 12 months after the last dose of rituximab. Men who are sexually active must use condoms during treatment period and 4 weeks after the last dose of any study drug.
6. Willing and able to participate in all required evaluations and procedures in this study protocol including swallowing capsules without difficulty.
7. Ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use protected health information.

Exclusion Criteria:

1. Diagnosed with mantle cell lymphoma
2. Previously treated with more than four lines of chemotherapy (Consolidative autologous stem cell transplantation is deemed as the same line therapy)
3. Previously treated with allogeneic hematopoietic stem cell transplantation within 6 months
4. GVHD requiring treatment
5. Patient who cannot take drug per oral
6. Known resistance to both BTK inhibitor and lenalidomide (Progression free survival to both BTK inhibitor and lenalidomide < 6 months)
7. Known resistant mutation to BTK inhibitor (BTKC481S and PLGCR665W)
8. Prior malignancy (or any other malignancy that requires active treatment), except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer from which the subject has been disease free for ≥ 5 years or which will not limit survival to < 5 years.
9. Clinically significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of screening, or any Class 3 or 4 cardiac disease as defined by the New York Heart Association Functional Classification. Subjects with controlled, asymptomatic atrial fibrillation during screening can enroll on study.
10. Malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel that is likely to affect absorption, symptomatic inflammatory bowel disease, partial or complete bowel obstruction, or gastric restrictions and bariatric surgery, such as gastric bypass.
11. Known history of infection with HIV or any uncontrolled active systemic infection (eg, bacterial, viral or fungal).
12. Known history of drug-specific hypersensitivity or anaphylaxis to study drug (including active product or excipient components).
13. Active bleeding, history of bleeding diathesis (eg, hemophilia or von Willebrand disease).
14. Uncontrolled AIHA (autoimmune hemolytic anemia) or ITP (idiopathic thrombocytopenic purpura).
15. Requires treatment with a strong cytochrome P450 3A4 (CYP3A4) inhibitor/inducer.
16. Requires or receiving anticoagulation with warfarin or equivalent vitamin K antagonists (eg, phenprocoumon) within 7 days of first dose of study drug.
17. Prothrombin time/INR or aPTT (in the absence of Lupus anticoagulant) > 2x ULN.
18. Requires treatment with proton pump inhibitors (eg, omeprazole, esomeprazole, lansoprazole, dexlansoprazole, rabeprazole, or pantoprazole). Subjects receiving proton pump inhibitors who switch to H2-receptor antagonists or antacids are eligible for enrollment to this study.
19. History of significant cerebrovascular disease or event, including stroke or intracranial hemorrhage, within 6 months before the first dose of study drug.
20. Major surgical procedure within 28 days of first dose of study drug. Note: If a subject had major surgery, they must have recovered adequately from any toxicity and/or complications from the intervention before the first dose of study drug.
21. Hepatitis B or C serologic status: subjects who are hepatitis B core antibody (anti-HBc) positive and who are surface antigen negative will need to have a negative polymerase chain reaction (PCR). Those who are hepatitis B surface antigen (HbsAg) positive or hepatitis B PCR positive will be excluded. Those who are positive only for anti-HBc and negative for HbsAg and hepatitis B PCR need to receive adequate antiviral prophylaxis for hepatitis B during the study period.

    Subjects who are hepatitis C antibody positive will need to have a negative PCR result. Those who are hepatitis C PCR positive will be excluded.
22. Active tuberculosis (history of exposure or history of positive tuberculin test; plus presence of clinical symptoms, physical or radiographic findings). Subjects with latent tuberculosis infection who are deemed to require treatment by the investigator are not eligible.
23. Uncontrolled active infection as determined by the investigator.
24. WBC < 3,000 /μL, ANC < 1,000 /μL, Platelets < 75,000 /μL, or Hemoglobin < 9.0 g/dL. Correction with transfusion within 2 weeks is not allowed.
25. Total bilirubin > 2 x ULN, or AST, ALT > 3 x ULN
26. Cr > 1.5 x ULN or CLcr < 30 mL/min/1.73m2
27. Breastfeeding or pregnant.
28. Concurrent participation in another therapeutic clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2019-07-09 (Actual); Primary Completion 2022-05-15 (Actual); Study Completion 2022-05-15 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | within 4 weeks after the 6 cycles of combination therapy (each cycle is 28 days)
  ORR is defined as the percentage of subjects with evidence of a confirmed complete response (CR) or partial response (PR) as per Lugano criteria

SECONDARY OUTCOMES:
Duration of response | Tumor status will be assessed at Week 8, 16, 24 (± 7 days), then every 3 months (± 14 days)
Complete remission rate | Response will be assessed at Week 8, 16, 24 (± 7 days)
Progression free survival | Tumor status will be assessed at Week 8, 16, 24 (± 7 days), then every 3 months (± 14 days)
Overall survival | Tumor status will be assessed at Week 8, 16, 24 (± 7 days), then every 3 months (± 14 days)

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Park C, Lee HS, Kang KW, Lee WS, Do YR, Kwak JY, Shin HJ, Kim SY, Yi JH, Lim SN, Lee JO, Yang DH, Jang H, Choi B, Lim J, Sun CH, Byun JM, Yoon SS, Koh Y. Combination of acalabrutinib with lenalidomide and rituximab in relapsed/refractory aggressive B-cell non-Hodgkin lymphoma: a single-arm phase II trial. Nat Commun. 2024 Mar 30;15(1):2776. doi: 10.1038/s41467-024-47198-4. PMID 38555311